CLINICAL TRIAL: NCT01676948
Title: An Open-label, Multi-arm, Non-comparative Safety and Tolerability Study of Canakinumab (ACZ885) in Patients With Active Systemic Juvenile Idiopathic Arthritis (SJIA)
Acronym: β-SPECIFIC 4Pa
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: PRINTO / PRCSG (Unknown)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CACZ885G2402; 2012-003054-92 (EudraCT Number)
Record Dates: First submitted 2012-08-29; First posted 2012-08-31 (Estimated); Last update posted 2015-10-15 (Estimated); Status verified 2015-10

CONDITIONS: Systemic Juvenile Idiopathic Arthritis
Keywords: SJIA; Systemic Juvenile Idiopathic Arthritis; children; systemic autoinflammatory disease, ACZ885, canakinumab; human monoclonal anti-interleukin-1β (IL-1 β) antibody; hildhood immunizations vaccinations
MeSH Terms: conditions — Arthritis, Juvenile | interventions — canakinumab

ARMS (6):
- Canakinumab - Cohort 1, 2mg (Experimental): 2 mg/kg q4wk (followed by taper to 1 mg/kg q4wk and drug discontinuation if appropriate)
  Interventions: Drug: Canakinumab
- Canakinumab - Cohort 1, 4mg (Experimental): 4 mg/kg q8wk (followed by taper to 4 mg/kg q12wk and drug discontinuation if appropriate)
  Interventions: Drug: Canakinumab
- Canakinumab - Cohort 2, 2mg (Experimental): 2 mg/kg q4wk (followed by taper to 1 mg/kg q4wk and drug discontinuation if appropriate)
  Interventions: Drug: Canakinumab
- Canakinumab - Cohort 2, 4mg (Experimental): 4 mg/kg q8wk (followed by taper to 4 mg/kg q12wk and drug discontinuation if appropriate)
  Interventions: Drug: Canakinumab
- Cohort 2 - canakinumab dose reduction (Experimental)
  Interventions: Drug: ACZ885
- Cohort 1 - canakinumab dose reduction (Experimental)
  Interventions: Drug: ACZ885

INTERVENTIONS:
Drug: ACZ885
  Arms: Cohort 1 - canakinumab dose reduction; Cohort 2 - canakinumab dose reduction
Drug: Canakinumab
  Arms: Canakinumab - Cohort 1, 2mg; Canakinumab - Cohort 1, 4mg
Drug: Canakinumab — Patients rolling over into this study from CACZ885G2301E1 (Cohort 1) will continue on their established canakinumab dose of either 4 mg/kg SC given every 4 weeks or 2mg/kg SC given every 4 weeks, until eligible for dose reduction.
  Canakinumab-naïve patients
  Arms: Canakinumab - Cohort 1, 2mg; Canakinumab - Cohort 2, 2mg
Drug: Canakinumab — Patients rolling over into this study from CACZ885G2301E1(Cohort 2) will receive a standard canakinumab dose of 4mg/kg SC given every 4 weeks, until eligible for dose reduction
  Arms: Canakinumab - Cohort 1, 2mg; Canakinumab - Cohort 1, 4mg; Canakinumab - Cohort 2, 2mg; Canakinumab - Cohort 2, 4mg

SUMMARY:
This two-part open-label, multi-arm, non-comparative study will collect long-term safety, efficacy and tolerability data from patients who were responsive to canakinumab from study CACZ885G2301E1 (Cohort 1), and from patients who are treatment naïve to canakinumab (Cohort 2). In addition, the effect of inactivated vaccines in an SJIA patient population will be assessed for the development of adequate (protective) antibody levels following immunization according to respective local vaccination guidelines.

Study Part I:

All patients will be treated with canakinumab 4 mg/kg every 4 weeks (or 2 mg/kg every 4 weeks for Cohort 1 patients who are receiving that dose in CACZ885G2301E1) until study end unless discontinuation occurs, or until they qualify for Part II of the study.

Study Part II:

Patients who are eligible will be randomized to receive canakinumab at a reduced dose or prolonged dose interval (see requirements for dose reduction/dose interval prolongation below).

Patients in Cohort 1 receiving 2 mg/kg q4wk in CACZ885G2301E1 will not be randomized but will be part of the treatment arm canakinumab dose reduction if they are eligible.

ELIGIBILITY:
Key inclusion criteria:

Cohort 1:

1. All patients currently enrolled in study CACZ885G2301E1, including patients who discontinued canakinumab therapy for inactive disease in CACZ885G2301E1 as per physician discretion and who are now currently in a flare and require canakinumab therapy again

Cohort 2:

1. Male and female patients aged ≥ 2 to < 20 years at the time of the screening visit
2. Confirmed diagnosis of SJIA as per ILAR definition that must have occurred at least 2 months prior to enrollment with an onset of disease < 16 years of age:

   • Arthritis in one or more joints, with or preceded by fever of at least 2 weeks duration that is documented to be daily/quotidian for at least 3 days and accompanied by one or more of the following:
   * Evanescent non-fixed erythematous rash,
   * Generalized lymph node enlargement,
   * Hepatomegaly and/ or splenomegaly,
   * Serositis
3. Active systemic disease at the time of baseline visit defined as having 2 or more of the following:

   * Documented spiking, intermittent fever (body temperature > 38°C) for at least 1 day during the screening period and within 1 week before first canakinumab dose,
   * At least 2 joints with active arthritis (using ACR definition of active joint),
   * C-reactive protein (CRP) > 30 mg/L (normal range < 10 mg/L),
   * Rash,
   * Serositis,
   * Lymphadenopathy,
   * Hepatosplenomegaly
4. Patient's willingness to discontinue anakinra, rilonacept, tocilizumab or other experimental drug under close monitoring
5. Patients who are scheduled to receive an immunization, according to their local vaccination guidelines, with an inactivated vaccine and willing to participate in the assessment schedule for vaccinated patients

Key exclusion criteria:

Cohort 1 and Cohort 2:

1. Active or recurrent bacterial, fungal or viral infection at the time of enrollment
2. Underlying metabolic, renal, hepatic, infectious or gastrointestinal conditions which in the opinion of the investigator immunocompromises the patient and/ or places the patient at unacceptable risk for participation in an immunomodulatory therapy.
3. History of malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases.
4. Live vaccinations within 3 months prior to the start of the study.

Cohort 2:

The following additional key exclusion criteria apply for Cohort 2.

1. Presence of moderate to severe impaired renal function
2. Clinical evidence of liver disease or liver injury as indicated by abnormal liver function tests at screening
3. History/evidence of macrophage activation syndrome within the previous 6 months

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 2 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2013-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Long-term safety and tolerability of canakinumab and the retention rate of canakinumab-treated patients | Days 1 to 533
  Outcome Measure Description: The long-term safety and tolerability of canakinumab and the retention rate of canakinumab-treated patients will be evaluated by monitoring of serious adverse events and adverse events leading to discontinuation of study drug.

SECONDARY OUTCOMES:
The percentage of patients who meet the adapted pediatric ACR, its individual components, and the Juvenile Arthritis Disease Activity Score [JADAS] over time | Days 1 to 533
  Outcome Measure Description: Patients will be classified into the adapted pediatric ACR categories to characterize their magnitude of efficacy response. JADAS will be derived from physician global assessment, parent/patient global assessment, active joint count and CRP.
The level of systemic corticosteroid tapering achieved in Part I | Day 1 to start of Part II
  Patients will be classified into the following 3 categories: ≥ 0.2 mg/kg at end of Part I, those who reach a corticosteroid dose between >0-<0.2 mg/kg and those who reach corticosteroid free regimen.
The level of canakinumab tapering achieved after randomization to the dose reduction arm or dose interval prolongation treatment arm in Part II | from start of Part II to Day 533
  In the canakinumab dose reduction arm, patients will be classified into the following 3 categories: Number of patients who are able to reach 1mg/kg q4wk at the end of Part II, canakinumab free regimen by the end of Part II and those who come back to 2mg/kg q4wk at the end of Part II.
  In the canakinumab dose interval arm, patients will be classified into the following 3 categories: Number of patients who are able to reach 4mg/kg q12wk at the end of Part II, canakinumab-free regimen by the end of Part II and those who come back to 4mg/kg q8wk at the end of Part II.
The time to treatment failure in Part II | from start of Part II to Day 533
  Time to treatment failure (TTF) is defined as time from randomization to the date when the patient's worsened SJIA disease activity requires increasing the doze or shortening the treatment interval of canakinumab or the date the patient is withdrawn from the study due to a safety concern.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals